CLINICAL TRIAL: NCT02294071
Title: Prospective Comparative Study of the Efficacy of Common Antipyretic Treatments in Febrile Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Rieder, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LHRI IRF
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Fever
Keywords: acetaminophen; ibuprofen
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- acetaminophen (Experimental): acetaminophen 15mg/kg (max 975mg)
  Interventions: Drug: Acetaminophen
- ibuprofen (Experimental): ibuprofen 10mg/kg (max 600mg)
  Interventions: Drug: Ibuprofen
- combination (Experimental): acetaminophen 15mg/kg (max 975mg) and ibuprofen 10mg/kg (max 600mg)
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — oral liquid ibuprofen 10mg/kg (maximum 600 mg)
  Other Names: Advil
  Arms: combination; ibuprofen
Drug: Acetaminophen — oral liquid acetaminophen 15mg/kg (max 975mg)
  Other Names: Tylenol
  Arms: acetaminophen; combination

SUMMARY:
This study will examine in detail the immediate effects of three common treatments given to children with fevers to lower their temperature. Each child will be given either ibuprofen, acetaminophen, or a combination, and their temperature monitored at five-minute intervals. The temperature-lowering effects of each treatment will be compared to evaluate which is most effective.

DETAILED DESCRIPTION:
There is no substantial evidence that a fever lower than 41°C is harmful to the welfare of an otherwise healthy child, although they can be dangerous to children already in critical condition [1,2]. However, fevers in healthy children commonly cause anxiety in parents and caregivers, so parents and physicians often give antipyretic medications to lower the fever [3,4]. Ibuprofen and acetaminophen are two of the most commonly used medications in children. Most major pediatric medical associations agree about appropriate dosages for children, but give no clear guidelines on whether ibuprofen or acetaminophen should be used [3,5]. Physicians commonly make the decision between the two based on their personal opinions of the efficacy and safety of the medications, or based on habit [6]. Survey data shows that more than half of physicians use combinations of both acetaminophen and ibuprofen to treat fever, either simultaneously or on an alternating schedule, with a variety of dosing patterns [6]. A majority of physicians believed there were established guidelines supporting this use, but in fact there are not [6].

Combining the two medications is widely theorized to improve effectiveness, but clinical trials comparing combination treatments to ibuprofen and/or acetaminophen alone have shown inconsistent results [4,7-12]. Several pharmacodynamic studies have shown that ibuprofen and acetaminophen both produce their largest effects on temperature within the first hour following dosage [9,10,13-16]. Despite this, only one study has been performed examining the change in temperature at intervals shorter than 30 minutes, and that study used substandard monitoring methods [10].

This study will use gold-standard monitoring methods to take temperatures every five minutes through the first one to four hours of treatment. Understanding the pattern of temperature change in the acute stages after dosing will help settle the debate about the optimal medication choice for treating childrens' fevers.

ELIGIBILITY:
Inclusion Criteria:

* fever between 38 and 41 Celsius (inclusive) on presentation to ER
* assessment by treating physician that patient requires antipyretic treatment

Exclusion Criteria:

* known allergy or hypersensitivity to either study medication
* received any antipyretic medication in past eight hours
* patient requires admission to hospital
* co-morbidities indicating increased risk of complication
* assessment by treating physician that patient is medically unsuitable for the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
temperature reduction from baseline | 4 hours
  change in temperature from baseline at time of drug administration and at five minute intervals afterward for a minimum of one hour, maximum 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rieder, MD, Principal Investigator — Western University, Canada

REFERENCES:
- [Background] Mullins ME, Empey M, Jaramillo D, Sosa S, Human T, Diringer MN. A prospective randomized study to evaluate the antipyretic effect of the combination of acetaminophen and ibuprofen in neurological ICU patients. Neurocrit Care. 2011 Dec;15(3):375-8. doi: 10.1007/s12028-011-9533-8. PMID 21503807
- [Background] Lee BH, Inui D, Suh GY, Kim JY, Kwon JY, Park J, Tada K, Tanaka K, Ietsugu K, Uehara K, Dote K, Tajimi K, Morita K, Matsuo K, Hoshino K, Hosokawa K, Lee KH, Lee KM, Takatori M, Nishimura M, Sanui M, Ito M, Egi M, Honda N, Okayama N, Shime N, Tsuruta R, Nogami S, Yoon SH, Fujitani S, Koh SO, Takeda S, Saito S, Hong SJ, Yamamoto T, Yokoyama T, Yamaguchi T, Nishiyama T, Igarashi T, Kakihana Y, Koh Y; Fever and Antipyretic in Critically ill patients Evaluation (FACE) Study Group. Association of body temperature and antipyretic treatments with mortality of critically ill patients with and without sepsis: multi-centered prospective observational study. Crit Care. 2012 Feb 28;16(1):R33. doi: 10.1186/cc11211. PMID 22373120
- [Background] Section on Clinical Pharmacology and Therapeutics; Committee on Drugs; Sullivan JE, Farrar HC. Fever and antipyretic use in children. Pediatrics. 2011 Mar;127(3):580-7. doi: 10.1542/peds.2010-3852. Epub 2011 Feb 28. PMID 21357332
- [Background] Wong T, Stang AS, Ganshorn H, Hartling L, Maconochie IK, Thomsen AM, Johnson DW. Combined and alternating paracetamol and ibuprofen therapy for febrile children. Cochrane Database Syst Rev. 2013 Oct 30;2013(10):CD009572. doi: 10.1002/14651858.CD009572.pub2. PMID 24174375
- [Background] D Leduc SWCPSCPC. Temperature measurement in pediatrics. Canadian Pediatric Society. 2013.
- [Background] Mayoral CE, Marino RV, Rosenfeld W, Greensher J. Alternating antipyretics: is this an alternative? Pediatrics. 2000 May;105(5):1009-12. doi: 10.1542/peds.105.5.1009. PMID 10790455
- [Background] Vyas FI, Rana DA, Patel PM, Patel VJ, Bhavsar RH. Randomized comparative trial of efficacy of paracetamol, ibuprofen and paracetamol-ibuprofen combination for treatment of febrile children. Perspect Clin Res. 2014 Jan;5(1):25-31. doi: 10.4103/2229-3485.124567. PMID 24551584
- [Background] Allan GM, Ivers N, Shevchuk Y. Treatment of pediatric fever: Are acetaminophen and ibuprofen equivalent? Can Fam Physician. 2010 Aug;56(8):773. No abstract available. PMID 20705883
- [Background] Erlewyn-Lajeunesse MD, Coppens K, Hunt LP, Chinnick PJ, Davies P, Higginson IM, Benger JR. Randomised controlled trial of combined paracetamol and ibuprofen for fever. Arch Dis Child. 2006 May;91(5):414-6. doi: 10.1136/adc.2005.087874. Epub 2006 Feb 7. PMID 16464962
- [Background] Hay AD, Costelloe C, Redmond NM, Montgomery AA, Fletcher M, Hollinghurst S, Peters TJ. Paracetamol plus ibuprofen for the treatment of fever in children (PITCH): randomised controlled trial. BMJ. 2008 Sep 2;337:a1302. doi: 10.1136/bmj.a1302. PMID 18765450
- [Background] Kramer LC, Richards PA, Thompson AM, Harper DP, Fairchok MP. Alternating antipyretics: antipyretic efficacy of acetaminophen versus acetaminophen alternated with ibuprofen in children. Clin Pediatr (Phila). 2008 Nov;47(9):907-11. doi: 10.1177/0009922808319967. Epub 2008 Jun 6. PMID 18539869
- [Background] Paul IM, Sturgis SA, Yang C, Engle L, Watts H, Berlin CM Jr. Efficacy of standard doses of Ibuprofen alone, alternating, and combined with acetaminophen for the treatment of febrile children. Clin Ther. 2010 Dec;32(14):2433-40. doi: 10.1016/j.clinthera.2011.01.006. PMID 21353111
- [Background] Brown RD, Kearns GL, Wilson JT. Integrated pharmacokinetic-pharmacodynamic model for acetaminophen, ibuprofen, and placebo antipyresis in children. J Pharmacokinet Biopharm. 1998 Oct;26(5):559-79. doi: 10.1023/a:1023225217108. PMID 10205771
- [Background] Kauffman RE, Sawyer LA, Scheinbaum ML. Antipyretic efficacy of ibuprofen vs acetaminophen. Am J Dis Child. 1992 May;146(5):622-5. doi: 10.1001/archpedi.1992.02160170102024. PMID 1621668
- [Background] Temple AR, Temple BR, Kuffner EK. Dosing and antipyretic efficacy of oral acetaminophen in children. Clin Ther. 2013 Sep;35(9):1361-75.e1-45. doi: 10.1016/j.clinthera.2013.06.022. Epub 2013 Aug 23. PMID 23972576
- [Background] Troconiz IF, Armenteros S, Planelles MV, Benitez J, Calvo R, Dominguez R. Pharmacokinetic-Pharmacodynamic Modelling of the antipyretic effect of two oral formulations of ibuprofen. Clin Pharmacokinet. 2000 Jun;38(6):505-18. doi: 10.2165/00003088-200038060-00004. PMID 10885587